CLINICAL TRIAL: NCT05814679
Title: The Effect of Relaxation With Virtual Reality on Fatigue and Comfort in Hemodialysis Patients
Brief Title: Relaxation With Virtual Reality on Fatigue and Comfort in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Neşe Altinok Ersoy, Research Assistant (pHD), Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E1-22-3047
Record Dates: First submitted 2023-03-07; First posted 2023-04-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The patient will relax with virtual reality in the hemodialysis center with the researcher.
  Interventions: Other: Relaxation with virtual reality
- Control Group (Placebo Comparator): The patients in the control group will be given a training on the functions of the kidneys.
  Interventions: Other: Attention match

INTERVENTIONS:
Other: Relaxation with virtual reality — In this research, a virtual reality relaxation video will be used in which the natural wonders are presented to the audience in an immersive environment.
  Arms: Intervention Group
Other: Attention match — kidney function instruction
  Arms: Control Group

SUMMARY:
Based on the task of providing the comfort of the patient, which is an indispensable part of the nursing profession, which many nurse theorists emphasize, there has been no study in the literature on the determination of the effect of virtual relaxation, which can be effective on the fatigue and comfort levels of patients receiving hemodialysis treatment. Therefore, the aim of this study is to examine the effect of virtual reality and relaxation on fatigue and comfort in hemodialysis patients.

DETAILED DESCRIPTION:
The patient will be prepared for relaxation with virtual reality and will be given a comfortable sitting position.

The patient will watch the relaxation practice with virtual reality once during the hemodialysis treatment.

The application will be terminated with the expiration of the virtual reality relaxation video.

Fatigue and comfort score will be measured after the application.

ELIGIBILITY:
Inclusion Criteria:

* Receiving hemodialysis treatment for the last 6 months
* Receiving four-hour hemodialysis treatment three times a week
* 18 years or older
* Deaf and visually impaired
* Without cognitive and psychiatric diagnosis
* Open to communication and cooperation
* Patients who agreed to participate in the study

Exclusion Criteria:

* Kidney transplant
* Discomfort due to virtual reality glasses
* Suspected/diagnosed COVID-19
* Patients who want to leave the study voluntarily
* Death

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | Assessing change of fatigue severity scale scores baseline, after each application for three weeks. Between third and fifth weeks any intervention will not be implemented and fatigue severity scale score will measure fifth week.
  In the study, fatigue symptom will be measured with the fatigue severity scale.
Hemodialysis Comfort Scale | Assessing change of fatigue comfort scale scores baseline, after each application for three weeks. Between third and fifth weeks any intervention will not be implemented and comfort scale score will measure fifth week.
  In the study, hemodialysis comfort will be measured with the hemodialysis comfort scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Cit Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No